CLINICAL TRIAL: NCT06684210
Title: Study of the Clinical Effect of External Oblique Muscle Intercostal Muscle Plane Block in Abdominal Surgery。
Brief Title: Study of the Clinical Effect of External Oblique Muscle Intercostal Muscle Plane Block in Abdominal Surgery
Acronym: EOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WCX123456
Record Dates: First submitted 2024-10-17; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Nerve Block; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External oblique intercostal plane block. (Experimental): Given 0.5% ropivacaine intercostal nerve block, 2.0ug/kg sufentanil + tropisetron 5mg intravenous analgesia.
  Interventions: Procedure: Intercostal plane block of the external oblique muscle
- Patient controlled in travenousanalgesia. (No Intervention): Given intravenous analgesia with 2.0ug/kg sufentanil + tropisetron 5 mg.

INTERVENTIONS:
Procedure: Intercostal plane block of the external oblique muscle — Under ultrasound guidance, a single dose of 0.25% ropivacaine 20ml was given for bilateral intercostal muscle plane block of external oblique muscles
  Arms: External oblique intercostal plane block.

SUMMARY:
This study intends to apply external oblique intercostal muscle plane block in thoracoabdominal resection, and to explore its effect on perioperative analgesia and rehabilitation quality in patients undergoing thoracoabdominal surgery.

DETAILED DESCRIPTION:
Approved by the hospital ethics committee, 60 patients undergoing thoracic and abdominal surgery were selected in this study. They were divided into experimental group (n=30) and control group (n=30). The experimental group was given 0.5% ropivacaine intercostal nerve block, 2.0ug/kg sufentanil and tropisetron 5mg intravenous analgesia, and the control group was given 2.0ug/kg sufentanil and tropisetron 5mg intravenous analgesia. MAP, HR and SPO2 were recorded at admission (T0), completion of induction (T1), skin incision (T2), 30min after operation (T3) and 30min after extubation (T5). The block range of nerve block in the experimental group was recorded. The VAS score and the number of patient-controlled analgesia pump were recorded 30min after extubation, 6h, 24h and 48h after operation in resting state and cough state. Postoperative adverse reactions such as respiratory depression, expectoration weakness, nausea, vomiting, and skin itching were recorded. The first time to get out of bed after operation was recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status Classification of I-II Aged 18-60 years old ; Will be scheduled to undergo elective LC

Exclusion Criteria:

* Coagulation disorders, Liver/kidney disease, Abdominal surgery history, Infection in the block application area, Chronic opioid use.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Patient's postoperative pain score | Extubation for 30minutes, 6 hours after surgery, 24 hours after surgery, and 48 hours after surgery
  Using the VIsual Analogue Scale,patients were guided to indicate the corresponding pain score according to their own pain situation, and the score ranged from 0 to 10. To evaluate the degree of postoperative pain, a score of 0 indicates no pain at all, a score of 2 indicates mild pain, and a score of 10 indicates the most severe pain, with higher scores indicating more severe pain

SECONDARY OUTCOMES:
Changes in blood pressure | Perioperative period
  Mean arterial pressure at different time points.Mean arterial pressure will be reported in mmHg.
Changes in heart rate | Perioperative period
  Heart rate at different time points.Heart rate will be reported in counts per minute.
Extent of action of external oblique intercostal muscle plane block | Ten minutes after the nerve block
  The specific extent of action of the external oblique muscle intercostal muscle plane block in the thoracoabdominal wall.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Qinhuangdao, Qinhuangdao, Hebei, China